CLINICAL TRIAL: NCT00588146
Title: Phase 2 Study of PEG-Intron in Hereditary Hemorrhagic Telangiectasia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Schering-Plough discontinued supplying study drug.
Sponsor: Mayo Clinic (Other)
Collaborators: Augusta University (Other); Unity Health Toronto (Other); Schering-Plough (Industry)
Responsible Party: Karen Swanson, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2400-05; R01FD003076-01 (FDA)
Record Dates: First submitted 2007-12-26; First posted 2008-01-08 (Estimated); Results first posted 2013-01-28 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Anemia; Liver Disease; Hypoxemia
Keywords: anemia; HHT; Liver disease; Hypoxemia; Iron deficiency anemia; Liver disease with high cardiac output; Diffuse pulmonary AVMs with hypoxemia
MeSH Terms: conditions — Anemia; Liver Diseases; Hypoxia; Anemia, Iron-Deficiency | interventions — peginterferon alfa-2b; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pegylated Interferon Alpha2b, then Standard Care (Experimental): Weekly subcutaneous injection of pegylated interferon alpha2b 1 microgram/kg/week for 6 months, then standard care for 6 months.
  Interventions: Drug: Pegylated Interferon Alpha2b; Other: Standard care
- Standard Care, then Pegylated Interferon Alpha2b (Experimental): Standard care for 6 months, then weekly subcutaneous injection of pegylated interferon alpha2b 1 microgram/kg/week for 6 months.
  Interventions: Drug: Pegylated Interferon Alpha2b; Other: Standard care

INTERVENTIONS:
Drug: Pegylated Interferon Alpha2b — Weekly subcutaneous injection of 1 microgram/kg/week
  Other Names: PEG-Intron
Other: Standard care — Standard care

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of pegylated interferon alpha-2b (PEG-Intron) in patients with severe complications related to Hereditary hemorrhagic telangiectasia (HHT).

Funding Source - FDA Office of Orphan Products Development (OOPD)

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety and tolerability of pegylated interferon alpha-2b (PEG-Intron) in patients with severe complications related to Hereditary Hemorrhagic Telangiectasia (HHT). Participants will be randomized to the treatment arm or control arm and then crossed over to the alternate arm at 6 months for the remainder of the 12-month study. Study treatment will consist of weekly subcutaneous injections of pegylated interferon alpha-2b (PEG-Intron), 1 microgram/kilogram/week. Adverse events as well as monitoring and treatment of toxicities will be followed as stated in the protocol. Adverse events will be graded according to the Modified NCI Common Toxicity Criteria. After every five participants have completed one month of treatment, an independent data safety monitoring board will review any adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Definite diagnosis of HHT by clinical criteria or genetic diagnosis. For the clinical diagnosis, 3 of the 4 following criteria1 must be present:

   1. Epistaxis: spontaneous, recurrent
   2. Telangiectases: multiple at characteristic sites
   3. Visceral lesions including telangiectases and/or arteriovenous malformations (AVM) (pulmonary, hepatic, gastrointestinal, cerebral, spinal)
   4. Family history of a first degree relative with HHT
2. Transfusion-dependent anemia from HHT-related bleeding (epistaxis from nasal mucosal telangiectases or gastrointestinal bleeding from gastrointestinal telangiectases) defined as a hemoglobin (Hb) < 9g/dL with transfusion of at least one unit of packed red blood cells within the past 6 months or Hb < 11g/dL in females or < 13g/dL in males with transfusion of at least 5 units of blood within the past 6 months. Patients must be on a stable dose of iron or intolerant of iron. Patients must have failed traditional treatment options.
3. Clinically stable outpatient
4. Able and willing to return for outpatient visits
5. Ability to perform subcutaneous injections
6. Adult (Age 18 - 70 years)
7. Presence of the following laboratory results at entry:

   1. White blood cell count ≥ 2000/mm^3
   2. Neutrophil count ≥ 1000/mm^3
   3. Platelet count ≥ 80,000/mm^3
   4. Thyroid stimulating hormone within normal limits (Minimal abnormalities of the sensitive thyroid stimulating hormone may be allowed provided that the free thyroxin is normal and the patient is clinically euthyroid)
8. Negative pregnancy test at enrollment, if applicable
9. If the participant is a sexually active woman of childbearing potential, evidence that she is practicing adequate contraception during the treatment period. Adequate contraception includes use of an intrauterine device, oral contraceptives, progesterone implanted rods, medroxyprogesterone acetate, surgical sterilization, barrier method (diaphragm + spermicide), a monogamous relationship with a male partner who has had a vasectomy or is using a condom + spermicide or a birth control method acceptable to the study physicians. Participants and/or their partners must agree to continue the use of adequate contraception for at least 6 months following completion of treatment.
10. Written informed consent specific for this protocol obtained prior to entry
11. Patients agree to take study medication as directed and follow all study related procedures until the conclusion of their protocol participation
12. Hepatic involvement by HHT characterized by high output heart failure due to hepatic vascular malformations (symptoms of heart failure including edema, ascites, S3 gallop, orthopnea, or jugular venous pressure > 10 cm H_2O) plus cardiac index (CI) measured at right heart catheterization > 4.4 L/min/m^2. Patients must have failed traditional treatment options.
13. Computed tomography scanning (CT) of the liver documenting vascular abnormalities consistent with HHT
14. Child-Pugh category A
15. Diffuse pulmonary telangiectases or AVMs documented by pulmonary angiography not amenable to treatment with embolization techniques. Patients must have failed traditional treatment options.
16. Positive contrast echocardiography documenting right to left intrapulmonary shunt
17. Resting or exercise-induced hypoxemia defined as a partial pressure of oxygen (PaO_2) < 70 mmHg at rest or an oxygen saturation (SpO_2) < 85% with exercise.

Exclusion Criteria:

1. Anemia from any other cause than that due to HHT-related bleeding
2. Hypersensitivity to PEG-Intron or any other component of the product
3. Decompensated liver disease

   1. Chronic active Hepatitis B infection
   2. Child-Pugh category B or C
4. History of severe psychiatric disease

   1. Prior suicide attempt
   2. Hospitalization for psychiatric disease
   3. Period of disability due to a psychiatric disease
   4. Current episode of moderate to severe depression not responsive to treatment
5. History of immunologically mediated disease

   1. Inflammatory bowel disease
   2. Idiopathic thrombocytopenic purpura
   3. Systemic lupus erythematosus
   4. Autoimmune hemolytic anemia
   5. Scleroderma
   6. Sarcoidosis
   7. Multiple sclerosis
   8. Severe psoriasis
   9. Clinical evidence of rheumatoid arthritis
   10. Autoimmune hepatitis
6. History of clinically significant cardiovascular disease

   1. Positive stress test
   2. Clinically significant arrhythmia
   3. Congestive heart failure
   4. Uncontrolled hypertension
   5. Coronary artery bypass surgery within 24 weeks prior to entry
   6. Angina pectoris or myocardial infarction within 1 year prior to entry
7. Seizure disorder uncontrolled by anticonvulsants (within the last 12 months)
8. History of thyroid disease poorly controlled on prescribed medications
9. History or evidence of retinopathy
10. Patients on chronic anticoagulation
11. History of chronic renal insufficiency (creatinine > 2.5 mg/dL)
12. Patients who have received an investigational drug within 24 weeks of treatment assignment
13. History or other evidence of severe illness or other comorbid condition which would make the patient unsuitable for participation in a research protocol
14. Liver dysfunction from any other cause than that due to HHT (chronic active hepatitis B infection, hepatitis C infection, alcoholic cirrhosis, etc.)
15. Cardiac index < 4.4 L/min/m^2
16. Pulmonary AVMs with feeding arteries > 3 mm in diameter amenable to embolization techniques
17. Other pulmonary diseases causing hypoxemia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Swanson, DO, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Mayo Clinic, Rochester, Minnesota from January 2007 through September 2010.
Period: First Intervention (Baseline to 6 mo)
Arm/Group | Pegylated Interferon Alpha2b, Then Standard Care | Standard Care, Then Pegylated Interferon Alpha2b
Started | 5 | 5
Completed | 1 | 2
Not Completed | 4 | 3
Not completed — Adverse Event | 4 | 3
Period: Second Intervention (6 Months to 1 Year)
Arm/Group | Pegylated Interferon Alpha2b, Then Standard Care | Standard Care, Then Pegylated Interferon Alpha2b
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to pegylated interferon alpha-2b first and standard care first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin
Description: The hemoglobin level is expressed as the amount of hemoglobin in grams (gm) per deciliter (dL) of whole blood.
Time Frame: baseline, one year
Population: Only 3 subjects completed the study, so the numbers were too low to analyze the study.
Arm/Group | Pegylated Interferon Alpha2b, Then Standard Care | Standard Care, Then Pegylated Interferon Alpha2b
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 1-year study by telephone or direct interview. Adverse events were graded according to Modified NCI Common Toxicity Criteria. If a subject discontinued for an adverse event, they were observed for 12 weeks.
Groups:
- Pegylated Interferon Alpha-2b: Weekly subcutaneous injection of pegylated interferon alpha2b 1 microgram/kg/week
- Standard Care: Subjects received standard care for hereditary hemorrhagic telangiectasia.
Arm/Group | Pegylated Interferon Alpha-2b | Standard Care
Serious Adverse Events (participants affected / at risk) | 3/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Interferon Alpha-2b (N=10) | Standard Care (N=10)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Interferon Alpha-2b (N=10) | Standard Care (N=10)
Seizure (General disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (2)
Myalgias (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthralgias (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Right flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early because Schering-Plough discontinued supplying study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No